CLINICAL TRIAL: NCT02315989
Title: A Study of the Early-Phase Safety of Proton Therapy Equipment for Patients Suffering From Solid Cancers, and the Equipment's Operational Effectiveness.
Brief Title: Early-Phase Safety of Proton Therapy Equipment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101-5215C
Record Dates: First submitted 2014-10-30; First posted 2014-12-12 (Estimated); Results first posted 2015-12-31 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2014-09

CONDITIONS: Malignant Glioma; Hepatocellular Carcinoma; Head and Neck Malignant Tumor; Prostate Cancer
MeSH Terms: conditions — Glioma; Carcinoma, Hepatocellular; Prostatic Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- safety (Other): proton therapy
  Interventions: Radiation: proton therapy

INTERVENTIONS:
Radiation: proton therapy — proton therapy

SUMMARY:
The main purpose of this study is to collect the safety data of Sumitomo Heavy Industries' proton therapy equipment for the treatment of solid cancer patients in Linkou Chang Gung Memorial Hospital, including the patients' early-stage adverse reactions and the efficacy on tumors, as well as to assess the operating functionality of the proton therapy system.

DETAILED DESCRIPTION:
The main purpose of this study is to collect the safety data of Sumitomo Heavy Industries' proton therapy equipment for the treatment of solid cancer patients in Linkou Chang Gung Memorial Hospital, including the patients' early-stage adverse reactions and the efficacy on tumors, as well as to assess the operating functionality of the proton therapy system.

In this study, solid cancer subjects will be treated with Sumitomo's proton therapy system. Safety and operating functionality data will be collected during the treatment and following-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are pathologically confirmed to be suffering from solid cancer or brain tumor
2. Subjects who are measurable or with disease that is evaluable
3. Subjects who are expected to survive for at least 90 days
4. Subjects who did not receive any treatment that may affect this treatment (such as PEI, TAE) 4 weeks before they are chosen to receive this treatment
5. ECOG Performance Status (ECOG PS): 0, 1 or 2
6. Patients who can cooperate with the treatment requirements and maintain the gestures required during the irradiation process
7. Patients with well functioning main organs
8. The subject retained main organ functions.
9. The subject age is between 20-75 years old

Exclusion Criteria:

1. Subjects who once received radiotherapy on the area planned to be irradiated
2. Subjects whose irradiated area has active or persistent infectious disease
3. Pregnant or possibly pregnant subjects
4. Subjects with other serious complications
5. Subjects who are judged by the Principle Investigator (or co-principle investigator) as unsuitable or because of other reasons described above
6. The subject has the radiotherapy contraindication
7. Breast feeding
8. All the subjects have no plan to conception during the treatment and within one year after treatment
9. Subject who has any electronic devices in the body which could be affected by radiotherapy and has chance to cause accident. For example: pacemaker, artificial heart, brain and spinal cord stimulation, semi-implantable and implantable electrical stimulation、artificial inner ear ...etc

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Hong Hong, Ph.D., Principal Investigator — Vice-President
Locations (1):
- ChangGungMH, Taoyuan District, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Safety
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Safety
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 61.5 [39 to 73]
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Rate and Severity of Adverse Reactions
Description: After enrollment, each patient has to receive physical examination, laboratory tests, and image studies as baseline. During the course of radiotherapy, patients will have weekly evaluations in physicals and laboratory tests. Image studies are optional during treatment. In the follow-up periods, monthly exams, including regular physicals, markers in serum and urine and image studies to evaluation treatment responses, will be scheduled till 90 days after the end of treatment.
Time Frame: Average 90 days after treatment.
Measure: Number; unit: participants
Arm/Group | Safety
Number analyzed (Participants) | 6
participants | 6

2. Secondary Outcome: Percentage of System Errors
Description: During treatment, the frequency of operation of the system error will be recorded and analyzed to see if the system can run smoothly.
Time Frame: Average 100 days after treatment.
Measure: Number; unit: percentage of system errors
Groups:
- The Frequency of Operation of the System Error: 6 subjects received a total of 165 proton therapy, a total of 21 times the system running abnormalities. There was no correlation between system abnormalities during the study and the adverse events.
Arm/Group | The Frequency of Operation of the System Error
Number analyzed (Participants) | 6
percentage of system errors | 12.7

3. Secondary Outcome: Percentage of Each Target Lesion Evaluation Types.(1)Complete Response(2)Partial Response,(3)Progressive Disease,(4)Stable Disease,(5) Inevaluable
Description: Response Evaluation Criteria In Solid Tumors:(1)complete Response(CR),Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm (2)Partial Response(PR), At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. (3)Progressive Disease(PD), At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (4)Stable Disease(SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. (5) Inevaluable (NE), Inevaluable for response: specify reasons (for example: early death, malignant disease; toxicity; tumor assessments not repeated/incomplete; other (specify).
Time Frame: Average 100 days after treatment.
Measure: Number; unit: percentage of participants
Groups:
- Stable Disease: Stable Disease(SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
- Partial Response: Partial Response(PR), At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
- Inevaluable: Inevaluable (NE), Inevaluable for response: specify reasons (for example: early death, malignant disease; toxicity; tumor assessments not repeated/incomplete; other (specify).
Arm/Group | Stable Disease | Partial Response | Inevaluable
Number analyzed (Participants) | 6 | 6 | 6
percentage of participants | 50 | 16.67 | 33.33

ADVERSE EVENTS:
Time Frame: 6 months (August, 2014-February, 2015)
Arm/Group | Safety
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety (N=6)
White blood cell decreased (Blood and lymphatic system disorders) | 1 — Case 1 On treatment: 1 Gr I "White blood cell decreased", 1 Gr II "White blood cell decreased"; Follow-up: 1 Gr I "White blood cell decreased"
Dermatitis radiation (Skin and subcutaneous tissue disorders) | 4 — Case 2 On treatment: 1 Gr I "Dermatitis radiation"; Case 4 On treatment: 1 Gr I & 1 Gr II "Dermatitis radiation"; Case 6 On treatment: 1 Gr I "Dermatitis radiation"; Case 7 On treatment: 2 Gr I & 1 Gr II "Dermatitis radiation";
Anal hemorrhage (Gastrointestinal disorders) | 1 — Case 3 On treatment: 1 Gr I "Anal hemorrhage", Follow-up: 1 Gr I "Anal hemorrhage",
Rectal hemorrhage (Gastrointestinal disorders) | 1 — Case 3 On treatment: 1 Gr II "Rectal hemorrhage",
Anemia (Blood and lymphatic system disorders) | 1 — Case 3 Follow-up: 1 Gr I "Anemia"
Alopecia (Skin and subcutaneous tissue disorders) | 1 — Case 4 On treatment: 1 Gr I "Alopecia",
Mucositis oral (Gastrointestinal disorders) | 2 — Case 6 On treatment: 2 Gr I & 1 Gr II "Mucositis oral" Case 7 On treatment: 2 Gr I & 1 Gr II "Mucositis oral"
Dysgeusia (Nervous system disorders) | 1 — Case 6 On treatment: 2 Gr I & 1 Gr II "Dysgeusia"; Follow-up: 1 Gr I "Dysgeusia",
Dysphagia (Gastrointestinal disorders) | 2 — Case 6 On treatment: 2 Gr I & 1 Gr II "Dysphagia" Case 7 On treatment: 2 Gr I & 1 Gr II "Dysphagia"
Dry mouth (Gastrointestinal disorders) | 2 — Case 6 On treatment: 1 Gr I & 1 Gr II "Dry mouth"; Follow-up: 1 Gr I "Dry mouth" Case 7 On treatment: 1 Gr I "Dry mouth"; Follow-up: 1 Gr I "Dry mouth"
Lip pain (Gastrointestinal disorders) | 2 — Case 6 On treatment: 1 Gr I & 1 Gr II "Lip pain", Case 7 On treatment: 2 Gr I & 1 Gr II "Lip pain"
Edema face (Gastrointestinal disorders) | 1 — Case 6 Follow-up: 1 Gr I "Edema face"
Trismus (Musculoskeletal and connective tissue disorders) | 1 — Case 7 On treatment: 1 Gr I "Trismus"; Follow-up: 1 Gr I "Trismus"
Constipation (Gastrointestinal disorders) | 1 — Case 7 On treatment: 1 Gr I "Constipation"

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No